CLINICAL TRIAL: NCT02812758
Title: Does Sedation Depth (as Evaluated by the Bispectral Index) Influence Dynamic Indices of Preload Dependence? An Observational, Single-centre Pilot Study
Brief Title: Does Sedation Depth (as Evaluated by the Bispectral Index) Influence Dynamic Indices of Preload Dependence?
Acronym: BIS2
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2015_843_0012
Record Dates: First submitted 2016-06-20; First posted 2016-06-24 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Thoracic Surgery
Keywords: sedation depth; indices of preload dependence
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- patients: All sedated, intubated, mechanically ventilated adult patients admitted for elective cardiac surgery, monitored for sedation depth (with the BIS) and for preload dependence indices (SVV, PPV and PVI) transthoracic echocardiography
  Interventions: Device: transthoracic echocardiography

INTERVENTIONS:
Device: transthoracic echocardiography — recording of data on cardiac output measured non-invasively by transthoracic echocardiography, including the SVV

SUMMARY:
Dynamic indices of preload dependence (such as stroke volume variability -SVV , pulse pressure variability - PPV and plethysmograph variability index - PVI ) are reportedly predictive of the response to vascular filling in sedated, mechanically ventilated patients. However, the influence of the sedation depth on these dynamic indices has never been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All sedated, intubated, mechanically ventilated adult (over-18) patients admitted for elective cardiac surgery, monitored for sedation depth (with the BIS) and for preload dependence indices (SVV, PPV and PVI)
* Good echogenicity
* Social security coverage

Exclusion Criteria:

* Pregnancy, legal guardianship
* Subjects with black skin (a known technical limitation of plethysmography)
* Cardiac arrhythmia
* Sepsis
* Poor echogenicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All sedated, intubated, mechanically ventilated adult (over-18) patients admitted for elective cardiac surgery, monitored for sedation depth (with the BIS) and for preload dependence indices (SVV, PPV and PVI)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-12; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Values of the dynamic indices (SVV, PPV and PVI) at different sedation levels (as evaluated by the BIS) | Day 0

SECONDARY OUTCOMES:
The proportion of patients that change their preload dependence status during a change in sedation depth (as evaluated by the BIS). | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel LORNE, Md, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France